CLINICAL TRIAL: NCT00808444
Title: Non-inferiority of a Commercial Lot of the Pneumococcal Vaccine GSK1024850A Compared to a Clinical Lot.
Brief Title: Primary Vaccination Study With a Pneumococcal Conjugate Vaccine in Healthy Children 6-12wks of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 111654
Record Dates: First submitted 2008-12-11; First posted 2008-12-15 (Estimated); Results first posted 2010-11-19 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2016-10

CONDITIONS: Infections, Streptococcal
Keywords: Pneumococcal vaccine; Immunogenicity; Primary vaccination; Safety; Pneumococcal disease
MeSH Terms: conditions — Streptococcal Infections; Pneumococcal Infections | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; DTPa-HBV-IPV combined vaccine; RIX4414 vaccine

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor

ARMS (2):
- Synflorix Clinical Lot & Infanrix Group (Experimental): Subjects received 3 doses of the clinical lot of Synflorix TM (GSK1024850A) intramuscularly in the right thigh at 2-3-5 months of age (= study month 0, 1, 3) co-administered with a DTPa-combined vaccine (Infanrix hexa TM (at 2, 3 and 5 months of age in Malaysia or 2 and 5 months of age in Singapore) or Infanrix-IPV/Hib TM (at 3 months of age in Singapore)) intramuscularly in the left thigh and Rotarix TM orally at 2-3 months of age (= study month 0, 1).
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A (different lots); Biological: Infanrix hexa; Biological: Infanrix-IPV/Hib; Biological: Rotarix
- Synflorix Commercial Lot Infanrix Group (Experimental): Subjects received 3 doses of the commercial lot of Synflorix TM (GSK1024850A) intramuscularly in the lright thigh at 2-3-5 months of age (= study month 0, 1, 3) co-administered with a DTPa-combined vaccine (Infanrix hexa TM (at 2, 3 or 5 months of age in Malaysia or 2 and 5 months in Singapore) or Infanrix-IPV/Hib TM (at 3 months of age in Singapore)) intramuscularly in the left thigh and Rotarix TM orally at 2-3 months of age (= study month 0, 1).
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A (different lots); Biological: Infanrix hexa; Biological: Infanrix-IPV/Hib; Biological: Rotarix

INTERVENTIONS:
Biological: Pneumococcal conjugate vaccine GSK1024850A (different lots) — Intramuscular injection, 3 doses
Biological: Infanrix hexa — Intramuscular injection, 3 doses in Malaysia and 2 doses in Singapore
  Other Names: DTPa-combined vaccine
Biological: Infanrix-IPV/Hib — Intramuscular injection, only for Visit 2 in Singapore
  Other Names: DTPa-combined vaccine
Biological: Rotarix — Oral, 2 doses
  Other Names: HRV vaccine

SUMMARY:
The purpose of the present study is to demonstrate that the changes in the manufacturing process for the commercial lot of the pneumococcal conjugate vaccine GSK1024850A have no clinical impact and that the immune responses are non-inferior to the immune responses induced by the clinical lot. The study will be conducted in Singapore and Malaysia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between, and including 6-12 weeks of age at the time of the first vaccination.
* Subjects for whom the investigator believes that their parent(s)/guardian(s) can and will comply with the requirements of the protocol.
* Written or oral, signed or thumb-printed informed consent obtained from the parent(s)/guardian(s) of the child/ward.
* Free of any known or suspected health problems (as established by medical history and clinical examination before entering into the study).
* Born after a gestation period of >= 36 to <= 42 weeks.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of the study vaccines, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth.
* A family history of congenital or hereditary immunodeficiency.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period (with the exception of hepatitis B immunoglobulins at birth).
* Previous vaccination against diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B, Haemophilus influenzae type b and/or Streptococcus pneumoniae (with the exception of vaccines where the first dose can be given within the first two weeks of life).
* Planned administration/administration of a vaccine not foreseen by the study protocol during the period starting 30 days before each dose of vaccine and ending 7 days after Dose 1 and Dose 2 and 30 days after Dose 3.
* History of, or intercurrent diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis, H. influenzae type b and rotavirus disease.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* History of any neurological disorders or seizures.
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrolment.
* Gastroenteritis within 7 days preceding the study vaccine administration.
* Any clinically significant history of chronic gastrointestinal disease including any uncorrected congenital malformation of the gastrointestinal tract, intussusception or other medical condition determined to be serious by the investigator.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 466 (Actual)
Dates: Start 2009-01-05; Primary Completion 2009-11-02 (Actual); Study Completion 2009-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Malaysia (2):
  - GSK Investigational Site, Kuala Lumpur
  - GSK Investigational Site, Seremban, Negeri Sembilan
- GSK Investigational Site, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Lim FS, Koh MT, Tan KK, Chan PC, Chong CY, Shung Yehudi YW, Teoh YL, Shafi F, Hezareh M, Swinnen K, Borys D. A randomised trial to evaluate the immunogenicity, reactogenicity, and safety of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) co-administered with routine childhood vaccines in Singapore and Malaysia. BMC Infect Dis. 2014 Oct 2;14:530. doi: 10.1186/1471-2334-14-530. PMID 25278086
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 111654 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111654 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111654 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111654 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111654 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111654 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111654 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Synflorix Commercial Lot & Infanrix Group: Subjects received 3 doses of the commercial lot of Synflorix TM (GSK1024850A) intramuscularly in the lright thigh at 2-3-5 months of age (= study month 0, 1, 3) co-administered with a DTPa-combined vaccine (Infanrix hexa TM (at 2, 3 or 5 months of age in Malaysia or 2 and 5 months in Singapore) or Infanrix-IPV/Hib TM (at 3 months of age in Singapore)) intramuscularly in the left thigh and Rotarix TM orally at 2-3 months of age (= study month 0, 1).
Period: Overall Study
Arm/Group | Synflorix Clinical Lot & Infanrix Group | Synflorix Commercial Lot & Infanrix Group
Started | 233 | 233
Completed | 232 | 232
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix Clinical Lot & Infanrix Group | Synflorix Commercial Lot & Infanrix Group | Total
Number analyzed (Participants) | 233 | 233 | 466
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 7.3 (1.35) | 7.2 (1.30) | 7.3 (1.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 104 | 217
  Male | 120 | 129 | 249

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of Antibodies Against Vaccine Components of the Pneumococcal Vaccine
Description: Concentrations are given as Geometric Mean Concentrations (GMCs) in microgram per milliliter (μg/mL).
  Vaccine pneumococcal serotypes assessed included 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F.
Time Frame: One month after primary immunization (month 4)
Population: Analysis was performed on the According-to-Protocol cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix Clinical Lot & Infanrix Group | Synflorix Commercial Lot & Infanrix Group
Number analyzed (Participants) | 219 | 218
μg/mL
  Anti-1 | 2.67 [2.46 to 2.91] | 2.46 [2.25 to 2.69]
  Anti-4 | 3.95 [3.59 to 4.36] | 3.14 [2.84 to 3.47]
  Anti-5 | 4.34 [3.95 to 4.76] | 3.59 [3.29 to 3.92]
  Anti-6B | 1.31 [1.16 to 1.48] | 1.23 [1.07 to 1.41]
  Anti-7: number analyzed (Participants) | 218 | 217
  Anti-7 | 3.10 [2.83 to 3.39] | 3.20 [2.92 to 3.51]
  Anti-9V | 3.34 [3.03 to 3.69] | 3.14 [2.83 to 3.49]
  Anti-14 | 5.13 [4.54 to 5.79] | 4.74 [4.23 to 5.32]
  Anti-18C | 5.00 [4.40 to 5.69] | 5.15 [4.43 to 5.97]
  Anti-19F | 6.69 [6.04 to 7.41] | 6.96 [6.26 to 7.73]
  Anti-23F | 1.98 [1.76 to 2.23] | 1.68 [1.49 to 1.90]

2. Primary Outcome: Concentration of Antibody Against Protein D (PD)
Description: Concentration was expressed as GMC in GSK's 22F enzyme-linked-immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: One month after primary immunization (month 4)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix Clinical Lot & Infanrix Group | Synflorix Commercial Lot & Infanrix Group
Number analyzed (Participants) | 219 | 218
EL.U/mL | 2543.6 [2319.4 to 2789.4] | 1869.8 [1671.2 to 2091.9]

3. Secondary Outcome: Number of Subjects With Anti-pneumococcal Vaccine Serotype Antibody Concentrations Equal to or Above 0.20 µg/mL
Description: Vaccine pneumococcal serotypes included 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F.
Time Frame: One month after primary immunization (month 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Clinical Lot & Infanrix Group | Synflorix Commercial Lot & Infanrix Group
Number analyzed (Participants) | 219 | 218
Participants
  Anti-1 | 219 | 218
  Anti-4 | 219 | 218
  Anti-5 | 218 | 218
  Anti-6B | 211 | 204
  Anti-7F: number analyzed (Participants) | 218 | 217
  Anti-7F | 218 | 217
  Anti-9V | 219 | 218
  Anti-14 | 218 | 218
  Anti-18C | 219 | 217
  Anti-19F | 218 | 217
  Anti-23F | 215 | 212

4. Secondary Outcome: Number of Subjects With Anti-pneumococcal Cross-reactive Serotype Concentrations Equal to or Above 0.20 µg/mL
Description: Anti-pneumococcal cross-reactive serotypes were 6A and 19A.
Time Frame: One month after primary immunization (month 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Clinical Lot & Infanrix Group | Synflorix Commercial Lot & Infanrix Group
Number analyzed (Participants) | 219 | 218
Participants
  Anti-6A | 152 | 132
  Anti-19A | 135 | 119

5. Secondary Outcome: Number of Subjects With Opsonophagocytic Activity Against Vaccine Pneumococcal Serotypes
Description: Vaccine pneumococcal serotypes included 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F, and 23F.
  Opsonophagocytic activity was defined as the dilution of serum (opsonic titer) able to sustain 50% killing of live pneumococci under the assay conditions. The cut-off of the assay was an opsonic titer equal to or greater than 8.
Time Frame: One month after primary immunization (month 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Clinical Lot & Infanrix Group | Synflorix Commercial Lot & Infanrix Group
Number analyzed (Participants) | 209 | 210
Participants
  Opsono-1 | 185 | 189
  Opsono-4: number analyzed (Participants) | 207 | 207
  Opsono-4 | 207 | 203
  Opsono-5: number analyzed (Participants) | 207 | 210
  Opsono-5 | 204 | 203
  Opsono-6B: number analyzed (Participants) | 205 | 206
  Opsono-6B | 196 | 191
  Opsono-7F: number analyzed (Participants) | 206 | 208
  Opsono-7F | 206 | 208
  Opsono-9V: number analyzed (Participants) | 207 | 208
  Opsono-9V | 207 | 208
  Opsono-14: number analyzed (Participants) | 209 | 208
  Opsono-14 | 208 | 207
  Opsono-18C: number analyzed (Participants) | 204 | 206
  Opsono-18C | 202 | 199
  Opsono-19F: number analyzed (Participants) | 206 | 206
  Opsono-19F | 202 | 200
  Opsono-23F: number analyzed (Participants) | 209 | 207
  Opsono-23F | 207 | 206

6. Secondary Outcome: Number of Subjects With Opsonophagocytic Activity Against Cross-reactive Pneumococcal Serotypes
Description: Cross-reactive pneumococcal serotypes were 6A and 19A.
  Opsonophagocytic activity was defined as the dilution of serum (opsonic titer) able to sustain 50% killing of live pneumococci under the assay conditions. The cut-off of the assay was an opsonic titer equal to or greater than 8.
Time Frame: One month after primary immunization (month 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Clinical Lot & Infanrix Group | Synflorix Commercial Lot & Infanrix Group
Number analyzed (Participants) | 197 | 200
Participants
  Opsono-6A | 173 | 171
  Opsono-19A: number analyzed (Participants) | 197 | 199
  Opsono-19A | 83 | 75

7. Secondary Outcome: Opsonophagocytic Titers of Cross-reactive Pneumococcal Serotypes
Description: Opsonophagocytic titers were expressed as GMTs.
  Cross-reactive pneumococcal serotypes included 6A and 19A.
Time Frame: One month after primary immunization (month 4)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Synflorix Clinical Lot & Infanrix Group | Synflorix Commercial Lot & Infanrix Group
Number analyzed (Participants) | 197 | 200
titer
  Opsono-6A | 230.8 [180.3 to 295.4] | 173.7 [133.9 to 225.3]
  Opsono-19A: number analyzed (Participants) | 197 | 199
  Opsono-19A | 18.1 [13.7 to 23.8] | 15.1 [11.5 to 19.8]

8. Secondary Outcome: Poliovirus Types 1, 2 and 3 Titers
Description: Titers were given as Geometric Mean Titers (GMTs).
Time Frame: One month after primary immunization (month 4)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Synflorix Clinical Lot & Infanrix Group | Synflorix Commercial Lot & Infanrix Group
Number analyzed (Participants) | 99 | 93
titer
  Anti-Polio 1 | 313.8 [250.4 to 393.3] | 328.7 [253.1 to 427.0]
  Anti-Polio 2: number analyzed (Participants) | 98 | 93
  Anti-Polio 2 | 278.7 [225.4 to 344.7] | 229.1 [176.9 to 296.6]
  Anti-Polio 3: number analyzed (Participants) | 97 | 93
  Anti-Polio 3 | 408.8 [330.1 to 506.4] | 449.4 [351.9 to 573.8]

9. Secondary Outcome: Concentrations of Antibodies Against Diphteria Toxoid (DT) and Tetanus Toxoid (TT)
Description: Concentrations were defined as GMCs in international units per milliter (IU/mL)
Time Frame: One month after primary immunization (month 4)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Synflorix Clinical Lot & Infanrix Group | Synflorix Commercial Lot & Infanrix Group
Number analyzed (Participants) | 109 | 107
IU/mL
  Anti-DT | 3.317 [2.895 to 3.800] | 3.353 [2.991 to 3.759]
  Anti-TT | 4.879 [4.358 to 5.502] | 4.476 [4.013 to 4.992]

10. Secondary Outcome: Concentration of Antibody Against Hepatitis B Surface Antigen (HBs) by Enzyme Linked ImmunoSorbent Assay (ELISA).
Description: Concentration was given as GMC in milli international units per milliliter (mIU/mL). As a decrease in the specificity of the anti-HB ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL), the table shows results following partial or complete reanalysis.
Time Frame: One month after primary immunization (month 4)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Synflorix Clinical Lot & Infanrix Group | Synflorix Commercial Lot & Infanrix Group
Number analyzed (Participants) | 87 | 97
mIU/mL | 1521.2 [1129.7 to 2048.4] | 2114.1 [1658.5 to 2694.9]

11. Secondary Outcome: Concentration of Antibody Against Rotavirus Immunoglobulin A (IgA)
Description: Concentration was expressed as GMC in units per milliliter (U/mL).
Time Frame: 3 months after primary immunization (month 4)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Synflorix Clinical Lot & Infanrix Group | Synflorix Commercial Lot & Infanrix Group
Number analyzed (Participants) | 105 | 106
U/mL | 141.1 [103.0 to 193.4] | 114.8 [85.0 to 155.1]

12. Secondary Outcome: Occurrence of Serious Adverse Events
Description: SAEs assessed include medical occurrences that result in death, is life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Following vaccination and throughout the entire study period (Month 0 to Month 4)
Population: Analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | Synflorix Clinical Lot & Infanrix Group | Synflorix Commercial Lot & Infanrix Group
Number analyzed (Participants) | 233 | 233
subjects | 18 | 7

13. Secondary Outcome: Opsonophagocytic Titers of Vaccine Pneumococcal Serotypes
Description: Titers are presented as Geometric Mean Titers (GMTs).
  Pneumococcal serotypes included 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F.
Time Frame: One month after primary immunization (month 4)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Synflorix Clinical Lot & Infanrix Group | Synflorix Commercial Lot & Infanrix Group
Number analyzed (Participants) | 209 | 210
titer
  Opsono-1 | 128.9 [102.7 to 161.7] | 122.1 [98.3 to 151.7]
  Opsono-4: number analyzed (Participants) | 207 | 207
  Opsono-4 | 698.3 [619.6 to 786.9] | 609.3 [519.6 to 714.3]
  Opsono-5: number analyzed (Participants) | 207 | 210
  Opsono-5 | 127.9 [109.0 to 149.9] | 98.6 [83.0 to 117.1]
  Opsono-6B: number analyzed (Participants) | 205 | 206
  Opsono-6B | 870.7 [710.2 to 1067.6] | 619.2 [483.4 to 793.2]
  Opsono-7F: number analyzed (Participants) | 206 | 208
  Opsono-7F | 3905.8 [3420.2 to 4460.4] | 3585.7 [3119.8 to 4121.2]
  Opsono-9V: number analyzed (Participants) | 207 | 208
  Opsono-9V | 1800.0 [1596.6 to 2029.3] | 1851.3 [1612.3 to 2125.8]
  Opsono-14: number analyzed (Participants) | 209 | 208
  Opsono-14 | 1521.0 [1313.3 to 1761.6] | 1485.8 [1280.5 to 1724.0]
  Opsono-18C: number analyzed (Participants) | 204 | 206
  Opsono-18C | 533.5 [461.8 to 616.4] | 383.9 [319.3 to 461.5]
  Opsono-19F: number analyzed (Participants) | 206 | 206
  Opsono-19F | 689.6 [581.1 to 818.2] | 573.5 [477.2 to 689.3]
  Opsono-23F: number analyzed (Participants) | 209 | 207
  Opsono-23F | 2716.7 [2316.3 to 3186.3] | 2379.5 [2043.4 to 2770.7]

14. Secondary Outcome: Number of Subjects With Solicited Local and General Symptoms.
Description: Solicited local symptoms were pain, redness and swelling.
  Solicited general symptoms were drowsiness, fever, irritability, loss of appetite, diarrhoea and vomiting.
Time Frame: Within 4 days (day 0-3) after vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, which inlcuded all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Clinical Lot & Infanrix Group | Synflorix Commercial Lot & Infanrix Group
Number analyzed (Participants) | 233 | 233
Participants
  Pain | 162 | 157
  Redness | 149 | 142
  Swelling | 133 | 124
  Drowsiness | 151 | 136
  Fever | 193 | 175
  Irritability | 168 | 171
  Loss of appetite | 127 | 121
  Diarrhoea | 53 | 54
  Vomiting | 44 | 46

15. Secondary Outcome: Concentrations of Antibodies Against Pertussis Toxoid (PT), Filamentous Haemagglutinin (FHA), Pertactin (PRN)
Description: Concentrations are expressed as GMCs in EL.U/mL.
Time Frame: One month after primary immunization (month 4)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix Clinical Lot & Infanrix Group | Synflorix Commercial Lot & Infanrix Group
Number analyzed (Participants) | 109 | 107
EL.U/mL
  Anti-PT | 46.5 [41.1 to 52.6] | 45.4 [39.8 to 51.7]
  Anti-FHA: number analyzed (Participants) | 107 | 107
  Anti-FHA | 179.2 [157.5 to 203.9] | 186.2 [165.5 to 209.5]
  Anti-PRN | 142.1 [123.2 to 164.0] | 128.3 [110.9 to 148.5]

16. Secondary Outcome: Concentration of Antibody Against Polyribosyl-ribitol Phosphate (PRP)
Description: Concentrain was expressed as GMC in µg/mL.
Time Frame: One month after primary immunization (month 4)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix Clinical Lot & Infanrix Group | Synflorix Commercial Lot & Infanrix Group
Number analyzed (Participants) | 112 | 108
µg/mL | 9.745 [7.807 to 12.164] | 6.387 [5.051 to 8.078]

17. Secondary Outcome: Occurrence of Unsolicited Adverse Events
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Within 31 days (day 0-30) after vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Clinical Lot & Infanrix Group | Synflorix Commercial Lot & Infanrix Group
Number analyzed (Participants) | 233 | 233
Participants | 88 | 96

ADVERSE EVENTS:
Time Frame: Frequent AEs were assessed during the 4-day (day 0-3) follow-up period after vaccination for solicited AEs and 31-day (day 0-30) follow-up period for unsolicited AEs. SAEs were assessed from month 0 until study end (month 4).
Arm/Group | Synflorix Clinical Lot & Infanrix Group | Synflorix Commercial Lot & Infanrix Group
Serious Adverse Events (participants affected / at risk) | 18/233 | 7/233
Other Adverse Events (participants affected / at risk) | 230/233 | 228/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix Clinical Lot & Infanrix Group (N=233) | Synflorix Commercial Lot & Infanrix Group (N=233)
Upper respiratory tract infection (Infections and infestations) | 5 | 0
Escherichia urinary tract infection (Infections and infestations) | 3 | 1
Gastroenteritis (Infections and infestations) | 4 | 0
Bronchiolitis (Infections and infestations) | 2 | 1
Head injury (Injury, poisoning and procedural complications) | 2 | 0
Kawasaki's disease (Vascular disorders) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Meningitis tuberculous (Infections and infestations) | 1 | 0
Meningitis viral (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0
Spinal muscular atrophy (Congenital, familial and genetic disorders) | 0 | 1
Vith nerve parlysis (Nervous system disorders) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix Clinical Lot & Infanrix Group (N=233) | Synflorix Commercial Lot & Infanrix Group (N=233)
Pain (General disorders) | 162 | 157
Redness (General disorders) | 149 | 142
Swelling (General disorders) | 133 | 124
Drowsiness (General disorders) | 151 | 136
Fever (General disorders) | 193 | 175
Irritability (General disorders) | 168 | 171
Diarrhoea (General disorders) | 53 | 54
Vomiting (General disorders) | 44 | 46
Upper respiratory tract infection (Infections and infestations) | 28 | 40
Loss of appetite (General disorders) | 127 | 121

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.